CLINICAL TRIAL: NCT05256992
Title: Impact Evaluation of the TYRO Champion Dads Project in Dallas, Texas
Brief Title: TYRO Champion Dads Project Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Anthem Strong Families (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/35
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fathers

STUDY DESIGN:
Intervention Model Description: Standard services delivered as primary services to participants in both study groups under a shared condition are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula. Optional services available to both study groups by selecting 1-3 hours of coursework from menu of courses that address a variety of needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-Enhanced Services (Standard + Ray of Hope) (Experimental): Treatment group participants receive standard and enhanced services. Standard services are delivered as primary services to participants in both study groups under a shared condition, and they are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula. Finally, only the treatment group receives 10 hours of the Ray of Hope curriculum as an enhanced service. Optional services are available to both study groups by selecting 1-3 hours of coursework from a menu of courses in the Mini-Clinic that address a variety of needs.
  Interventions: Other: Standard Servies + Ray of Hope Curriculum; Other: Standard Services
- Control-Standard Services (Experimental): Only standard services are delivered to participants in the control group under a shared condition with the treatment group, and they are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula. Optional services are available to both study groups by selecting 1-3 hours of coursework from a menu of courses that address a variety of needs.
  Interventions: Other: Standard Services

INTERVENTIONS:
Other: Standard Servies + Ray of Hope Curriculum — Standard services delivered as primary services to participants in both study groups under a shared condition are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula. Optional services available to both study groups by selecting 1-3 hours of coursework from menu of courses that address a variety of needs.
  Arms: Treatment-Enhanced Services (Standard + Ray of Hope)
Other: Standard Services — Standard services delivered as primary services to participants in both study groups under a shared condition are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula.

SUMMARY:
This impact evaluation aims to determine if the addition of 10 hours of domestic violence prevention programming is effective at improving outcomes among those program participants who are randomly assigned to the treatment group. Both study groups will receive standard TYRO Champion Dads services (the TYRO Dads and TYRO Core Communication evidence-based curricula, plus support services), but only the treatment group will be offered the additional Ray of Hope curriculum hours focused on mitigating risk factors related to domestic violence.

DETAILED DESCRIPTION:
Anthem Strong Families (ASF) is reviewing the Ray of Hope curriculum as a possible addition to standard TCD services to better meet the needs of populations that may have unmet needs to address domestic violence in their families. The Ray of Hope curriculum is designed to help participants develop communication and conflict management skills like Core Communication but is a more robust approach since it adds a sharp focus on the dynamics of domestic violence and related risk factors.

The impact of the addition of the Ray of Hope curriculum will be assessed by comparing outcomes for participants who receive standard TYRO Champion Dads (TCD) services, which includes the TYRO curriculum plus support services, and participants who receive both standard services plus 10 Ray of Hope curriculum hours.

Goal 1: determine if treatment group participants who receive enhanced TCD services report healthier parenting attitudes compared to control group participants who receive only standard TCD services 6 months after TCD enrollment.

Goal 2: determine if treatment group participants who receive enhanced TCD services report healthier partner relationship behavior compared to control group participants who receive only standard TCD services 6 months after TCD enrollment.

Goal 3: determine if treatment group participants who receive enhanced TCD services report healthier parenting behavior compared to control group participants who receive only standard TCD services 6 months after TCD enrollment.

Goal 4: determine if treatment group participants who receive enhanced TCD services report healthier co-parenting behavior compared to control group participants who receive only standard TCD services 6 months after TCD enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Father (children must be no more than 24 years of age)
* must have no open criminal cases (can be deferred)

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father
* Has an open criminal case

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a fatherhood grant. Fathers or father-figures are accepted into the study.
Enrollment: 748 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Anthem Strong Families, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Started | 382 | 366
Completed | 382 | 366
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services | Total
Number analyzed (Participants) | 382 | 366 | 748
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 377 | 361 | 738
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 37.92 [19 to 73] | 37.72 [18 to 70] | 37.82 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 379 | 365 | 744
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 11 | 18
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 139 | 103 | 242
  White | 155 | 153 | 308
  More than one race | 75 | 95 | 170
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measures 1: Healthy Parenting Behavior
Description: What is the impact of enhanced TCD services (treatment) compared to standard TCD services only (control) on healthy parent behavior 6 months after TCD enrollment?
  * Average of 11 survey items that relate to frequency of positive interactions with participant's youngest child using categories on a five-point scale where 1 is never and 5 is every day or almost every day
  * Higher scores are always positive
  The 11 items are measured as a construct. All items are added together and divided by 11 to create the construct score.
  maximum score of 5.0, minimum score of 1.0
Time Frame: change from baseline to 6-months after enrollment
Population: There was a low number of participants who responded to this item in the final analysis in both the baseline and the follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Number analyzed (Participants) | 34 | 26
score on a scale | 3.88 (0.871) | 3.67 (1.017)

2. Primary Outcome: Primary Outcome Measures 2: Healthy Parenting Behavior
Description: What is the impact of enhanced TCD services (treatment) compared to standard TCD services only (control) on healthy parent behavior 6 months after TCD enrollment?
  • 1 survey item measures the reported frequency of fighting with their child on a five-point scale where 1 is never and 5 is every day or almost every day
  o A lower score is better
  maximum score of 5.0, minimum score of 1.0
Time Frame: baseline to 6-months after enrollment
Population: A low number of participants responded to this item on both the baseline and follow-up.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Number analyzed (Participants) | 52 | 40
score on scale | 4.5 (0.776) | 4.74 (0.554)

3. Primary Outcome: Primary Outcome Measure 3: Healthy Co-parenting Behavior
Description: What is the impact of enhanced TCD services (treatment) compared to standard TCD services only (control) on healthy co-parent behavior 6 months after TCD enrollment?
  • 11 survey items measure the reported frequency of agreement with key co-parenting behaviors using categories on a 5-point scale (1 'Strongly Disagree', 2 'Disagree', 3 'Neither Agree Nor Disagree', 4 'Agree', 5 'Strongly Agree').
  The 11 items are measured as a construct. All items are added together and divided by 11 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: change from baseline to 6-months after enrollment
Population: A low number of participants responded to this item on both the baseline and follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Number analyzed (Participants) | 34 | 40
score on a scale | 3.51 (0.593) | 3.50 (0.444)

4. Primary Outcome: Primary Outcome Measures 4: Healthy Partner Relationship Behavior
Description: • Average of 8 survey items related to frequency of disagreement with partner on different topics using categories on a 5-point scale where 1 is never and 5 is always
  Lower scores are positive and show a better outcome.
  The 8 items are measured as a construct. All items are added together and divided by 8 to create the construct score.
  maximum score of 5.0, minimum score of 1.0
Time Frame: change from baseline to 6-months after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Number analyzed (Participants) | 143 | 123
score on a scale | 3.94 (1.027) | 3.97 (0.901)

5. Secondary Outcome: Secondary Outcome Measure 1: Healthy Parenting Attitudes
Description: What is the impact of enhanced TCD services (treatment) compared to standard TCD services only (control) on healthy parenting attitudes 6-months after TCD enrollment?
  • 7 survey items measure the reported frequency of healthy parenting attitudes using categories on a 5-point scale (1 'Always', 2 'Often', 3 'Rarely', 4 'Sometimes', 5 'Never').
  The 7 items are measured as a construct. All items are added together and divided by 7 to create the construct score. The lower the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: baseline to 6-months after enrollment
Population: A low number of participants responded to this item on both the baseline and follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
Number analyzed (Participants) | 12 | 18
score on a scale | 4.72 (0.337) | 4.76 (0.392)

ADVERSE EVENTS:
Time Frame: 6-months through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Treatment-Enhanced Services (Standard + Ray of Hope) | Control-Standard Services
All-Cause Mortality (participants affected / at risk) | 0/382 | 0/366
Serious Adverse Events (participants affected / at risk) | 0/382 | 0/366
Other Adverse Events (participants affected / at risk) | 0/382 | 0/366

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT05256992/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT05256992/SAP_001.pdf